CLINICAL TRIAL: NCT07206381
Title: EMDR Group Therapy for Earthquake-Exposed Trauma Survivors: A Randomized Trial of Psychological and QEEG Outcomes
Brief Title: Effects of EMDR on Psychological Symptoms and EEG Findings in Trauma-Exposed Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Galata University (Other)
Responsible Party: Principal Investigator, Çiğdem Kınık, Assistant Professor, Istanbul Galata University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMDR-EEG-TR-2025
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: PTSD - Post Traumatic Stress Disorder; Depression; Anxiety Disorders and Symptoms; Sleep Quality; Quality of Life
Keywords: Eye Movement Desensitization and Reprocessing (EMDR); Posttraumatic Stress Disorder (PTSD); Depression; Anxiety; Sleep quality; quality of life; earthquake; QEEG
MeSH Terms: conditions — Combat Disorders; Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing; Psychotherapy, Group

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in parallel to either an EMDR intervention group or a waitlist control group. The EMDR group will receive 5-7 sessions of standardized group therapy, while the control group will not receive any intervention during the study period but will be offered EMDR after study completion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR Group (Experimental): Participants will receive 5-7 sessions of Eye Movement Desensitization and Reprocessing (EMDR) group therapy, delivered face-to-face by trained therapists, in line with the standard EMDR protocol. EEG measurements and psychological scales will be administered before and after the intervention.
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing (EMDR) Group Therapy
- Waitlist Control (No Intervention): Participants in this arm will not receive any active psychotherapy intervention during the study period. They will undergo baseline and post-test EEG recordings and psychological assessments at the same time intervals as the experimental group. For ethical reasons, they will be offered EMDR therapy after the study is completed if requested.

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing (EMDR) Group Therapy — Sessions conducted in groups with one therapist and one co-therapist; each session follows the EMDR standard protocol.
  Arms: EMDR Group

SUMMARY:
This study will examine the effects of Eye Movement Desensitization and Reprocessing (EMDR) group therapy on adults who experienced the April 2025 Silivri earthquake in Turkey. Participants will be randomly assigned to either an EMDR intervention group or a waitlist control group. Psychological symptoms will be measured using the PTSD Checklist for DSM-5 (PCL-5), the Depression, Anxiety, and Stress Scale (DASS-21), the Short Form Health Survey (SF-36), and the Pittsburgh Sleep Quality Index (PSQI). Quantitative EEG (QEEG) recordings will also be collected before and after the intervention to assess changes in brain activity related to emotional regulation and trauma processing. The goal of the study is to evaluate whether EMDR produces both clinical and neurophysiological improvements in trauma-exposed individuals.

DETAILED DESCRIPTION:
Traumatic experiences often lead to persistent psychological symptoms such as posttraumatic stress, depression, anxiety, and sleep disturbances, which significantly impair quality of life. Eye Movement Desensitization and Reprocessing (EMDR) is an evidence-based intervention for trauma-related disorders, and growing evidence suggests that it may also produce measurable changes in brain activity. This randomized controlled trial will evaluate the effects of EMDR group therapy on both clinical outcomes and neurophysiological markers in adults exposed to the April 2025 Silivri earthquake in Turkey.

Forty participants meeting inclusion criteria will be randomly assigned to either an EMDR intervention group (20 participants) or a waitlist control group (20 participants). The intervention group will receive 5-7 sessions of standardized EMDR group therapy, delivered face-to-face by trained therapists. Quantitative EEG (QEEG) recordings will be collected at baseline and after the intervention to assess changes in spectral power, frontal alpha asymmetry, and coherence patterns. Clinical outcomes will be measured with validated self-report instruments assessing PTSD symptoms, depression, anxiety, stress, sleep quality, and overall health-related quality of life.

This study is designed to test the hypothesis that EMDR group therapy produces significant improvements in both psychological symptoms and EEG biomarkers compared to a waitlist control. By integrating subjective self-report and objective neurophysiological data, the trial aims to provide a comprehensive evaluation of EMDR's therapeutic effects in trauma-exposed populations.

ELIGIBILITY:
Inclusion Criteria:

* Meeting DSM-5 criteria for posttraumatic stress symptoms following the April 2025 Silivri earthquake
* Age between 18 and 50 years
* Either medication-free for at least 1 month or on a stable dose of psychotropic medication
* No medical contraindications for EEG recording (e.g., no epilepsy, no metal implants)

Exclusion Criteria:

* Current diagnosis of schizophrenia, bipolar disorder, or a neurological disorder
* Receiving psychotherapy
* Inability to attend sessions regularly due to logistical or cognitive limitations

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-04 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in Posttraumatic Stress Symptoms (PCL-5) | Baseline (Pre-intervention, T1; Week 0) and Post-intervention (T2; Week 6, after completion of EMDR intervention)
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report scale measuring the severity of posttraumatic stress disorder symptoms according to DSM-5 criteria. Scores range from 0 to 80, with higher scores indicating more severe PTSD symptoms. Change in total score from baseline (pre-intervention) to post-intervention will be assessed.
Change in Quantitative EEG (QEEG) Power Spectral Measures | Baseline (Pre-intervention, T1; Week 0) and Post-intervention (T2; Week 6, after completion of EMDR intervention)
  EEG recordings will be collected using the Neuron-Spectrum-5 device according to the international 10-20 system. Power spectral analyses will be performed across frequency bands (delta, theta, alpha, beta, high beta). Changes in absolute and relative power from baseline to post-intervention will be examined.

SECONDARY OUTCOMES:
Change in Quality of Life (SF-36) | Baseline (Pre-intervention, T1; Week 0) and Post-intervention (T2; Week 6, after completion of EMDR intervention)
  The Short Form Health Survey (SF-36) is a 36-item measure of health-related quality of life, covering physical functioning, role limitations, pain, general health, vitality, social functioning, and emotional well-being. Scores range from 0 to 100, with higher scores reflecting better quality of life. Change in domain scores will be assessed from baseline to post-intervention.
Change in Depression, Anxiety, and Stress (DASS-21) | Baseline (Pre-intervention, T1; Week 0) and Post-intervention (T2; Week 6, after completion of EMDR intervention)
  The Depression, Anxiety, and Stress Scale-21 (DASS-21) is a 21-item self-report instrument measuring emotional distress across three subscales (depression, anxiety, stress). Scores range from 0 to 42 for each subscale, with higher scores indicating greater severity. Change in scores will be assessed from baseline to post-intervention.
Change in Sleep Quality (PSQI) | Baseline (Pre-intervention, T1; Week 0) and Post-intervention (T2; Week 6, after completion of EMDR intervention)
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item self-report questionnaire assessing sleep quality and disturbances over the past month. Scores range from 0 to 21, with higher scores indicating poorer sleep quality. Change in total score will be assessed from baseline to post-intervention.

IPD SHARING:
Plan to Share IPD: No
De-identified EEG data and questionnaire scores will be shared upon reasonable request after study completion, in compliance with ethical approval.

REFERENCES:
- [Background] Colvonen PJ, Glassman LH, Crocker LD, Buttner MM, Orff H, Schiehser DM, Norman SB, Afari N. Pretreatment biomarkers predicting PTSD psychotherapy outcomes: A systematic review. Neurosci Biobehav Rev. 2017 Apr;75:140-156. doi: 10.1016/j.neubiorev.2017.01.027. Epub 2017 Jan 28. PMID 28143760
- [Background] van der Kolk BA, Spinazzola J, Blaustein ME, Hopper JW, Hopper EK, Korn DL, Simpson WB. A randomized clinical trial of eye movement desensitization and reprocessing (EMDR), fluoxetine, and pill placebo in the treatment of posttraumatic stress disorder: treatment effects and long-term maintenance. J Clin Psychiatry. 2007 Jan;68(1):37-46. doi: 10.4088/jcp.v68n0105. PMID 17284128
- [Background] Jokic-Begic N, Begic D. Quantitative electroencephalogram (qEEG) in combat veterans with post-traumatic stress disorder (PTSD). Nord J Psychiatry. 2003;57(5):351-5. doi: 10.1080/08039480310002688. PMID 14522608
- [Background] Butt M, Espinal E, Aupperle RL, Nikulina V, Stewart JL. The Electrical Aftermath: Brain Signals of Posttraumatic Stress Disorder Filtered Through a Clinical Lens. Front Psychiatry. 2019 May 31;10:368. doi: 10.3389/fpsyt.2019.00368. eCollection 2019. PMID 31214058
- [Background] Pagani M, Di Lorenzo G, Verardo AR, Nicolais G, Monaco L, Lauretti G, Russo R, Niolu C, Ammaniti M, Fernandez I, Siracusano A. Neurobiological correlates of EMDR monitoring - an EEG study. PLoS One. 2012;7(9):e45753. doi: 10.1371/journal.pone.0045753. Epub 2012 Sep 26. PMID 23049852
- [Background] Pagani M, Di Lorenzo G, Monaco L, Daverio A, Giannoudas I, La Porta P, Verardo AR, Niolu C, Fernandez I, Siracusano A. Neurobiological response to EMDR therapy in clients with different psychological traumas. Front Psychol. 2015 Oct 27;6:1614. doi: 10.3389/fpsyg.2015.01614. eCollection 2015. PMID 26579006
- See also: ORCID profile of Principal Investigator — https://orcid.org/0009-0000-5236-2968